CLINICAL TRIAL: NCT05551767
Title: Induction Immunochemotherapy in Stage III-IVa Cancer of Oropharynx, Hypopharynx and Larynx
Brief Title: Induction Immunochemotherapy in Stage III-IVa Head and Neck Cancer
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: City Clinical Oncology Hospital No 1 (Other Government)
Collaborators: Moscow City Oncology Hospital No. 62 (Other Government); Moscow Clinical Scientific Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HN01
Record Dates: First submitted 2022-09-16; First posted 2022-09-23 (Actual); Last update posted 2022-09-23 (Actual); Status verified 2022-09

CONDITIONS: Neck Cancer
MeSH Terms: conditions — Head and Neck Neoplasms | interventions — pembrolizumab; Cisplatin; Fluorouracil

STUDY DESIGN:
Intervention Model Description: 3 cycles of induction immunochemotherapy with platinum (cisplatin 75 mg\m2, 5-FU 1000 mg/m2/day 96-hour infusion and pembrolizumab 200 mg) followed by (chemo)radiation.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Experimental arm (Experimental): 3 cycles of induction immunochemotherapy with platinum (cisplatin 75 mg\m2, 5-FU 1000 mg/m2/day 96-hour infusion and pembrolizumab 200 mg) followed by (chemo)radiation. Effect of induction therapy will be assesed by PET/CT and by endoscopic evaluation with biopsy of suspected residual tumor. Managemant of any residual tumor will be performed according with local rules and standards.
  Interventions: Drug: Pembrolizumab

INTERVENTIONS:
Drug: Pembrolizumab — 3 cycles of induction immunochemotherapy with platinum (cisplatin 75 mg\m2, 5-FU 1000 mg/m2/day 96-hour infusion and pembrolizumab 200 mg)
  Other Names: cisplatin and 5-FU

SUMMARY:
patients with locally advanced cancer of oropharynx, hypopharynx or larynx and CPS>1 will recieve 3 cycles of induction immunochemotherapy with platinum, 5-FU and pembrolizumab followed by (chemo)radiation.

DETAILED DESCRIPTION:
patients with locally advanced cancer of oropharynx, hypopharynx or larynx and CPS>1 will recieve 3 cycles of induction immunochemotherapy with platinum (cisplatin 75 mg\m2, 5-FU 1000 mg/m2/day 96-hour infusion and pembrolizumab 200 mg) followed by (chemo)radiation. Effect of induction therapy will be assesed by PET/CT and by endoscopic evaluation with biopsy of suspected residual tumor. Managemant of any residual tumor will be performed according with local rules and standards.

ELIGIBILITY:
Inclusion Criteria:

* Squamous cell cancer of oropharynx (p16+: T0-3N3, T4N0-3, p16- : T3-4aN0-1, T1-4aN2-3), hypopharynx (T2-3N0-3, T1N+, T4aN0-3) or larynx III-IVa (T1-2N2-3, T3N2-3, T4aN0-3) , TNM8 staging classification;
* Tumor is morphlogically confirmed;
* CPS>1 (22C3 clone);
* ECOG 0-2;
* Age above 18 years;
* Signed Informed consent form.

Exclusion Criteria:

* Cancer of nasopharynx;
* Non-squamous cell carcimomas or absense of morphological confirmation of squamous cell cancer;
* Stages I or II;
* ECOG>=3.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2022-08-30 (Actual); Primary Completion 2023-12-30 (Estimated); Study Completion 2024-12-30 (Estimated)

PRIMARY OUTCOMES:
complete response rate | through study completion, an average of 3 years
  rate of patients with no residual tumor after induction therapy including chemotherapy and radiotherapy
progression-free survival | through study completion, an average of 3 years
  Time from start of treatment to radiological disease progression

SECONDARY OUTCOMES:
overall survival | through study completion, an average of 3 years
  Time from start of treatment to death from any case
objective response rate | through study completion, an average of 3 years
  response rate by RESCIST 1.1
Organ-preserving treatment rate | through study completion, an average of 3 years
  rate of patients with organ sparing treatment

CONTACTS AND LOCATIONS:
Overall Officials: Vsevolod N Galkin, Professor, Principal Investigator — City Clinical Oncology Hospital No 1
Locations (3):
- Russia (3):
  - Moscow Clinical Scientific Center named after Loginov, Moscow
  - City clinical oncology hospital 1, Moscow
  - Moscow City Oncology Hospital No 62, Moscow

IPD SHARING:
Plan to Share IPD: No